CLINICAL TRIAL: NCT01297153
Title: Aphakia vs Pseudophakia - Randomized Clinical Trial in Children Under 2 Years Undergoing Bilateral Congenital Cataract Surgery
Brief Title: Aphakia Versus Pseudophakia in Children Under 2 Years Undergoing Bilateral Congenital Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Dr. Abhay R. Vasavada, Iladevi Cataract & IOL Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: icircAP
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Congenital Cataract
Keywords: Congenital Cataract; Children younger than 2 years; Aphakia; Primary IOL Implantation
MeSH Terms: conditions — Aphakia | interventions — Lenses, Intraocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aphakia (Active Comparator): * The patient is randomly assigned for aphakia / pseudophakia. This is done only after vitrectomy. If it is aphakia,IOL will not be implanted.Aphakia will be corrected with aphakic glasses / contact lenses. Bilateral aphakes are given both contact lenses and glasses. So when they do not wear contact lenses they can put on aphakic glasses. Unilateral aphakes are given only contact lenses. Contact lenses should be fitted in the eye in OT immediately after the operation.
  * Aphakic glasses :
  Prescribed within 2 weeks of surgery for both eyes.
  Interventions: Device: No IOL
- Pseudophakia (Active Comparator): The patient is randomly assigned for aphakia / pseudophakia. This is done only after vitrectomy. Hydrophobic Acrysof IOL is implanted.All pseudophakic children will be refracted and given the residual correction within a month of surgery.
  Interventions: Device: Intraocular Lens (Acrysof IOL)

INTERVENTIONS:
Device: Intraocular Lens (Acrysof IOL) — IOL fixation, material and size are important determinants of immediate and long-term outcome. In-the-bag fixation is the most preferred site of IOL implantation.
  Other Names: Hydrophobic Acrylic IOL
  Arms: Pseudophakia
Device: No IOL — No IOL will be implanted in these eyes
  Arms: Aphakia

SUMMARY:
The purpose of this study is to document the safety and efficacy of primary IOL implantation in children below 2 years of age undergoing congenital cataract surgery.

DETAILED DESCRIPTION:
The use of IOLs in pediatric patients has become increasingly popular in recent years and may represent a standard of care for older children. The refinements in surgical techniques attained in adult cataract surgery have been translated to pediatric cataract surgery to produce a technically safe eye. Nevertheless, the use of IOLs in children younger than 2 years remains controversial. Exaggerated inflammation, capsular opacification and changing refractive status of the developing eye should be considered before the use of IOLs in the first two years of life. Further more, there is concern about the unknown risks of an IOL over the long life span.

Currently, there are 3 methods of optical rehabilitation following congenital cataract surgery :

1. Primary IOL implantation.
2. Aphakic glasses.
3. Contact lenses.

At present, there is no randomized clinical trial reported to document the safety and efficacy of IOL implantation in children less than 2 years.

Aim : To compare the technical outcome (safety) and functional outcome (benefits) following primary IOL implantation and aphakia in children less than 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 2 years
* Congenital cataract
* Bilateral cataracts
* IOL fixation - Bag/Ciliary fixated

Exclusion Criteria:

* Microphthalmos (Mean axial length 2 SDs less than normal for age)
* Microcornea (Horizontal corneal diameter <9.5 mm-asper that particular age)
* Iris coloboma
* PHPV
* Aniridia
* *Glaucoma - IOP more than or equal to 25 mmHg

  * One eyed
  * Cataract surgery already performed in fellow eye

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2003-05; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Visual axis obscuration | 4 years
  Visual axis obscuration(VAO) assesed on slitlamp or under operating microscope in dilated pupil.VAO is defined as fibrous or proliferative cell growth leadind to a dull retinoscopic reflex.
Glaucoma | 4 years
  Intraocular pressure (IOP) measured with Perkins handheld applanation tonometer.
  Glaucoma defined as :
  IOP>21 mmHg >1 occasion with any of these 3 criteria
  1. Optic nerve cupping asymmetry >0.2 cd ratio asymmetry , CD ratio >0.4
  2. Abnormal asymmetrical axial length elongation
  3. Corneal oedema or enlargement
Central Corneal Thickness | 4 Years
  Corneal thickness assessed by ultrasonic pachymetry. An average of 3 values with an error less than 0.001 would be taken into account.

SECONDARY OUTCOMES:
Visual Acuity | 4 years .
  An Objective visual assessment to be performed using Lea Grating Paddles(Grating Acuity Test developed by Lea Hyvarinen16), Cardiff Acuity Cards(Preferential Looking Test17), or ETDRS (Early Treatment of Diabetic Retinopathy Study) chart. Vision is subjectively assessed as the ability to follow or to fixate on a point source of light or on an object shown to the child.. Ocular alignment was measured using alternative cover testing. If this kind of testing was not feasible, Hirschberg testing was performed..

CONTACTS AND LOCATIONS:
Overall Officials: Abhay R Vasavada, MS,FRCS, Principal Investigator — Iladevi Cataract And IOL Research Centre
Locations (1):
- Iladevi Cataract & IOL Research Centre, Ahmedabad, India